CLINICAL TRIAL: NCT03937375
Title: Re-Evaluation of the Effects of High PEEP During General Anesthesia For Surgery - An Individual Patient Data Meta-Analysis of PROVHILO, iPROVE and PROBESE
Brief Title: Re-Evaluation of the Effects of High PEEP During General Anesthesia For Surgery (REPEAT)
Acronym: REPEAT
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Hospital Carl Gustav Carus (Other); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: REPEAT
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2019-04

CONDITIONS: Surgery; Mechanical Ventilation Complication; Pulmonary Complication
Keywords: Surgery; Mechanical ventilation; PEEP; Postoperative pulmonary complications; Individual patient data meta-analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High PEEP: Use of high levels of PEEP with recruitment maneuvers
  Interventions: Behavioral: High PEEP
- Low PEEP: Use of low levels of PEEP without recruitment maneuvers
  Interventions: Behavioral: Low PEEP

INTERVENTIONS:
Behavioral: High PEEP — Use of high levels of PEEP combined with recruitment maneuvers and low tidal volume ventilation during general anesthesia
  Groups: High PEEP
Behavioral: Low PEEP — Use of low levels of PEEP without recruitment maneuvers and low tidal volume ventilation during general anesthesia
  Groups: Low PEEP

SUMMARY:
Aiming to understand the isolated impact of high PEEP in patients undergoing mechanical ventilation for general anesthesia for surgery, three appropriately sized international multicentre randomized controlled trials have been performed over recent years: the 'PROtective Ventilation using HIgh versus LOw PEEP trial (PROVHILO), the 'individualized PeRioperative Open-lung Ventilation trial' (iPROVE), and the 'Protective intraoperative ventilation with higher versus lower levels of positive end-expiratory pressure in obese patients trial' (PROBESE). These three trials had several similarities in key areas of their study protocols, inclusion and exclusion criteria, and collected data, and even the primary and secondary outcomes. Of note, the three trials combined high PEEP with recruitment manoeuvres. This allows an individual patient data meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

- Enrolled into one of the three studies (PROVHILO, iPROVE or PROBESE) to either high PEEP or low PEEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mechanical ventilation for general anesthesia for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3837 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications | Until day seven or hospital discharge, whichever comes first
  Collapsed composite of complications developing within the first seven postoperative days, including: Mild respiratory failure; or Severe respiratory failure; or Acute Respiratory Distress Syndrome (ARDS); or Pulmonary infection; or Pleural effusion; or Atelectasis; or Pneumothorax; or Bronchospasm.

SECONDARY OUTCOMES:
Incidence of severe postoperative pulmonary complications | Until day seven or hospital discharge, whichever comes first
  Collapsed composite of complications developing within the first seven postoperative days, including: Severe respiratory failure; or Acute Respiratory Distress Syndrome (ARDS); or Pulmonary infection; or Pleural effusion; or Atelectasis; or Pneumothorax; or Bronchospasm
Incidence of extrapulmonary pulmonary complications | Until day seven or hospital discharge, whichever comes first
  Collapsed composite of complications developing within the first seven postoperative days, including: Systemic Response Inflammatory Syndrome; or Sepsis; or Septic Shock; or Acute Kidney Injury.
Incidence of intraoperative complications | Intraoperatively
  Defined as intraoperative hypotension; or need for rescue for desaturations; or need for vasoactive drugs.
Incidence of intensive care unit admission | Until hospital discharge, death or 100 days, whichever comes first
  Incidence of intensive care unit admission during hospital stay
Hospital length of stay | Until hospital discharge, death or 100 days, whichever comes first
  Duration of hospital length of stay in days
Incidence of 7-day mortality | Until day seven or hospital discharge, whichever comes first
  Mortality during the first seven days of hospitalization
Incidence of in-hospital mortality | Until hospital discharge, death or 100 days, whichever comes first
  Mortality during hospitalization
Incidence of major postoperative complications | Until day seven or hospital discharge, whichever comes first
  Collapsed composite of complications developing within the first seven postoperative combining severe postoperative pulmonary complications, sepsis, septic shock and/or acute kidney injury)

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Germany
- Amsterdam UMC, University of Amsterdam, Amsterdam, Netherlands
- Hospital Clinico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The harmonized dataset will be available after the publication of the main results and under request to the steering committee
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After the publication of the main results

REFERENCES:
- [Background] Hemmes SN, Severgnini P, Jaber S, Canet J, Wrigge H, Hiesmayr M, Tschernko EM, Hollmann MW, Binnekade JM, Hedenstierna G, Putensen C, de Abreu MG, Pelosi P, Schultz MJ. Rationale and study design of PROVHILO - a worldwide multicenter randomized controlled trial on protective ventilation during general anesthesia for open abdominal surgery. Trials. 2011 May 6;12:111. doi: 10.1186/1745-6215-12-111. PMID 21548927
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Ferrando C, Soro M, Canet J, Unzueta MC, Suarez F, Librero J, Peiro S, Llombart A, Delgado C, Leon I, Rovira L, Ramasco F, Granell M, Aldecoa C, Diaz O, Balust J, Garutti I, de la Matta M, Pensado A, Gonzalez R, Duran ME, Gallego L, Del Valle SG, Redondo FJ, Diaz P, Pestana D, Rodriguez A, Aguirre J, Garcia JM, Garcia J, Espinosa E, Charco P, Navarro J, Rodriguez C, Tusman G, Belda FJ; iPROVE investigators (Appendices 1 and 2). Rationale and study design for an individualized perioperative open lung ventilatory strategy (iPROVE): study protocol for a randomized controlled trial. Trials. 2015 Apr 27;16:193. doi: 10.1186/s13063-015-0694-1. PMID 25927183
- [Background] Ferrando C, Soro M, Unzueta C, Suarez-Sipmann F, Canet J, Librero J, Pozo N, Peiro S, Llombart A, Leon I, India I, Aldecoa C, Diaz-Cambronero O, Pestana D, Redondo FJ, Garutti I, Balust J, Garcia JI, Ibanez M, Granell M, Rodriguez A, Gallego L, de la Matta M, Gonzalez R, Brunelli A, Garcia J, Rovira L, Barrios F, Torres V, Hernandez S, Gracia E, Gine M, Garcia M, Garcia N, Miguel L, Sanchez S, Pineiro P, Pujol R, Garcia-Del-Valle S, Valdivia J, Hernandez MJ, Padron O, Colas A, Puig J, Azparren G, Tusman G, Villar J, Belda J; Individualized PeRioperative Open-lung VEntilation (iPROVE) Network. Individualised perioperative open-lung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med. 2018 Mar;6(3):193-203. doi: 10.1016/S2213-2600(18)30024-9. Epub 2018 Jan 19. PMID 29371130
- [Background] Bluth T, Teichmann R, Kiss T, Bobek I, Canet J, Cinnella G, De Baerdemaeker L, Gregoretti C, Hedenstierna G, Hemmes SN, Hiesmayr M, Hollmann MW, Jaber S, Laffey JG, Licker MJ, Markstaller K, Matot I, Muller G, Mills GH, Mulier JP, Putensen C, Rossaint R, Schmitt J, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE investigators; PROtective VEntilation Network (PROVEnet); Clinical Trial Network of the European Society of Anaesthesiology (ESA). Protective intraoperative ventilation with higher versus lower levels of positive end-expiratory pressure in obese patients (PROBESE): study protocol for a randomized controlled trial. Trials. 2017 Apr 28;18(1):202. doi: 10.1186/s13063-017-1929-0. PMID 28454590
- [Derived] Serpa Neto A, Campos NS, Bluth T, Hemmes SNT, Ferrando C, Librero J, Soro M, Ball L, Mazzinari G, de Abreu MG, Schultz MJ; for REPEAT on behalf of the PROVHILO , iPROVE and PROBESE Investigators, and the PROVE Network investigators. Win Ratio approach for the composite outcome of postoperative pulmonary complications: Secondary analysis of a harmonised and pooled database of three randomised clinical trials. Eur J Anaesthesiol. 2025 Apr 1;42(4):340-346. doi: 10.1097/EJA.0000000000002116. Epub 2024 Dec 18. PMID 39698861
- [Derived] Mazzinari G, Zampieri FG, Ball L, Campos NS, Bluth T, Hemmes SNT, Ferrando C, Librero J, Soro M, Pelosi P, Gama de Abreu M, Schultz MJ, Serpa Neto A; PROVHILO investigators; iPROVE investigators; PROBESE investigators; PROVE network investigators. Effect of intraoperative PEEP with recruitment maneuvers on the occurrence of postoperative pulmonary complications during general anesthesia--protocol for Bayesian analysis of three randomized clinical trials of intraoperative ventilation. F1000Res. 2023 Jun 23;11:1090. doi: 10.12688/f1000research.125861.2. eCollection 2022. PMID 37234075
- [Derived] Campos NS, Bluth T, Hemmes SNT, Librero J, Pozo N, Ferrando C, Ball L, Mazzinari G, Pelosi P, Gama de Abreu M, Schultz MJ, Serpa Neto A; REPEAT; investigators for the PROVHILO study; iPROVE study; PROBESE study investigators; PROVE Network. Intraoperative positive end-expiratory pressure and postoperative pulmonary complications: a patient-level meta-analysis of three randomised clinical trials. Br J Anaesth. 2022 Jun;128(6):1040-1051. doi: 10.1016/j.bja.2022.02.039. Epub 2022 Apr 15. PMID 35431038

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03937375/Prot_SAP_000.pdf